CLINICAL TRIAL: NCT00194090
Title: A Double-blind, Placebo-controlled, Crossover Pilot Study of the Efficacy of Celecoxib 200 mg qd in Relieving Pain and Walking Dysfunction in Osteoarthritis of the Knee
Brief Title: Efficacy of Celecoxib vs Placebo to Prevent Pain in a Paced Walk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-04-41
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
Keywords: pain; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
A paced 20-minute walk is a reproducible model for acute pain in knee osteoarthritis

DETAILED DESCRIPTION:
This is a randomizd, placbo-controlled, crossover trial comparing a single dose of celecoxib to placebo measuring the time to onset of acute pain in a paced 20-minute walk.

40 subjects will be enrolled

ELIGIBILITY:
Inclusion Criteria:

Knee osteoarthritis by ACR clinical criteria Pain of at least 40 mm by VAS at baseline

-

Exclusion Criteria:

Non-pregant, non-lactating Able to stop active arthritis medication for washout Cardiovascular risk factors Abnormal EKG -

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2005-09-01 (Actual); Study Completion 2005-09-01 (Actual)

PRIMARY OUTCOMES:
time to onset of severe pain

SECONDARY OUTCOMES:
time to onset of moderate pain

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Hooper, MD, MS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- See also: hospital site to inquire about clinical trials — http://www.uhhs.com